CLINICAL TRIAL: NCT06545565
Title: Prevention of Metabolic Acidosis in Preterm Neonates by Replacing Sodium Chloride With Sodium Acetate in Parenteral Nutrition - A Randomized Controlled Trial. (PROTECT Trial)
Brief Title: Prevention of Metabolic Acidosis in Preterm Neonates by Replacing Sodium Chloride With Sodium Acetate in Parenteral Nutrition
Acronym: PROTECT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, Adnan Mirza, Clinical Assistant Professor, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024-6523-29448
Record Dates: First submitted 2024-07-30; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Metabolic Acidosis; Neonatal Disease; Neonatal Complication
Keywords: metabolic acidosis; sodium acetate; neonates; Parenteral Nutrition
MeSH Terms: conditions — Acidosis; Infant, Newborn, Diseases; Hyperphagia | interventions — Sodium Acetate; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Infants who will meet the inclusion criteria and whose parents will consent to participate will be randomized to one of the two intervention groups (So-A, or the standard So-C) prior to the preparation and commencement of PN. Randomization will be performed by pharmacists at the Sterile Preparation/Parenteral Unit of AKU hospital upon enrolment of each case. The randomization process will be performed according to a computer-generated list. For multiple births, each infant will be individually randomized.
  The interventional group: This group will receive sodium acetate in the neonatal PN.
  Control Group: The control group will receive sodium chloride in the neonatal PN.
  Intervention of the study: Use of sodium acetate in neonatal PN.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sodium acetate (Experimental)
  Interventions: Drug: sodium acetate group will receive sodium acetate in the neonatal PN.
- Sodium Chloride (Active Comparator)
  Interventions: Drug: sodium chloride group will receive sodium chloride in the neonatal PN.

INTERVENTIONS:
Drug: sodium acetate group will receive sodium acetate in the neonatal PN. — This group will receive sterile sodium acetate daily in the neonatal PN for the duration the patient will receive parenteral nutrition, a maximum of 28 days of life.
  Other Names: Sodium Acetate
  Arms: sodium acetate
Drug: sodium chloride group will receive sodium chloride in the neonatal PN. — This group will receive sterile sodium chloride daily in the neonatal PN for the duration the patient will receive parenteral nutrition, a maximum of 28 days of life.
  Other Names: sodium Chloride
  Arms: Sodium Chloride

SUMMARY:
The goal of this clinical trial is to learn if the addition of sodium acetate in neonatal PN works to prevent and treat metabolic acidosis and associated comorbidities in preterm neonates. It will also teach about the optimal doses of sodium acetate in PN. The main questions it aims to answer are:

Is the incidence of metabolic acidosis reduced in preterm neonates who received daily Sodium acetate in PN therapy (treatment) during the initial weeks of life compared with individuals who received sodium chloride in PN (standard)? Is the rate of neonatal comorbidities reduced in preterm neonates who received daily Sodium acetate in PN therapy (treatment) during the initial weeks of life compared with individuals who received sodium chloride in PN (standard)? What are the optimal neonatal dosing recommendations/guidelines of sodium acetate in daily PN, which are required to prevent/treat metabolic acidosis in the early life of preterm neonates? Researchers will compare Sodium acetate in PN therapy to sodium chloride in PN to see if Sodium acetate works to prevent and treat metabolic acidosis and associated comorbidities.

Included Participants:

All the neonates were admitted to the NICU of AKUH and received PN during 28 days of their lives.

Participants will receive sodium acetate or sodium chloride Written informed consent was obtained by parents/legal representatives (according to local regulations) before the initiation of PN. Gestational age < 33 weeks Included in the study before 72 hours of life

DETAILED DESCRIPTION:
Background Providing optimal nutritional support to extremely preterm and very low birth weight (VLBW) infants is still very much a challenge, as enteral feeding is generally delayed due to the prematurity of gastrointestinal function; these infants have poor sucking and swallowing reflexes, and there are concerns that a liberal feeding strategy may lead to complications, such as feeding intolerance or necrotizing enterocolitis (NEC). Early nutritional support is primarily delivered through parenteral nutrition (PN) is essential in the critical management during the neonatal period in these preterm babies.

PN provides all the required nutritional needs of preterm, including fluid, calories, and electrolytes. Sodium is both an electrolyte and a mineral. It helps keep the water (the amount of fluid inside and outside the body's cells) and electrolyte balance of the body. Sodium is also important in how nerves and muscles work. Most of the sodium in the body (about 85%) is found in blood and lymph fluid. Sodium is also provided through PN in two forms The first form is sodium chloride. In most parts of the world, sodium supplementation in PN has largely been in the form of sodium chloride. This is also the standard of care in the neonatal intensive care unit of Aga Khan University Hospital. Sodium chloride is added to the PN according to the sodium levels and body fluid balance.

The second source of sodium is sodium acetate, which is new in Aga Khan University Hospital but internationally used in PN. Daily sodium acetate will be added to the PN bag according to the sodium levels, acid-base balance, and total fluid intake. With the addition of sodium acetate, neonates have fewer metabolic acidosis complications, are more effective in preventing comorbidities, and are being used in the NICUs of developed countries.

MATERIALS AND METHODS Design This will be a 2-arm open-label phase III randomized controlled trial (RCT) to compare Sodium acetate and Sodium chloride, given daily as the component of parenteral nutrition over during first 28 days of life. Investigators will initiate the treatment within the first 72 hours following birth.

Setting This study will be conducted in the Neonatal Intensive Care Unit (NICU) of the Aga Khan University Hospital (AKUH), which is a 700-bedded, not-for-profit tertiary care hospital receiving country-wide referrals.

The interventional group: This group will receive sodium acetate in the neonatal PN.

Control Group: The control group will receive sodium chloride in the neonatal PN.

Intervention of the study: Use of sodium acetate in neonatal PN.

Data collection:

All relevant maternal and infant demographic data/Baseline characteristics, blood investigation results, and clinical outcomes will be recorded prospectively. The primary outcomes, pH, and base excess (BE) will be recorded from pre-PN on the first day of life (DOL), then 2- 7 DOL, and days 10, 13, 16,20,25, and 28 of life. For infants requiring less than 28 days of hospital stay, data will be collected till discharge/death.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained by parents/legal representative (according to local regulations) before the initiation of PN.
2. All the neonates who were admitted to the NICU of AKUH and received PN during 28 days of their life.
3. Gestational age < 33 weeks

Exclusion Criteria:

1. Infants with an inborn error of metabolism
2. Genetic or congenital condition that affects neurodevelopment or requires multiple surgeries (e.g., congenital viral infection, hydrops, complex congenital heart disease, severe dysmorphic features, etc.)
3. Severe metabolic alkalosis, in critically ill neonates, is defined as a persistent elevation of the serum pH above 7.45 and it also involves a primary increase in serum bicarbonate (HCO3-) concentration > 25mEq/L.
4. Severe Hypernatremia, in critically ill neonates, is defined as persistently high serum sodium levels > 150 mmol/L
5. Severe liver failure and syndromic infants with multiple congenital abnormalities and severe perinatal asphyxia

   -

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-05-10 (Estimated)

PRIMARY OUTCOMES:
metabolic acidosis | Blood-ph and serum-bicarbonate concentration will be recorded from pre-PN on the first day of life (DOL), then 2-7 DOL, and days 10,13,16,20,25&28 of life. For infants requiring <28 days of hospital stay until discharge/death.
  Severe metabolic acidosis, in critically ill neonates, is defined as a persistent low Blood pH < 7.26 and it also involves a primary decrease in serum bicarbonate (HCO3-) concentration <16 mEq/L]

SECONDARY OUTCOMES:
Development of Comorbid conditions (Bronchopulmonary dysplasia (BPD), patent ductus arteriosus (PDA), Intraventricular hemorrhage (IVH), Retinopathy of prematurity (ROP), necrotizing enterocolitis (NEC), Sepsis and jaundice ). | From the date of randomization until the date of first documented comorbid condition, assessed up to 28 days of life or date of death from any cause, whichever came first.
Duration of ventilation | Participants will be assessed from the date of randomization up to 28 days of life or date of death from any cause, whichever came first.
  number of days participant receive ventilatory support
Weight change (gain/loss) | Participants will be assessed for daily weight from the date of randomization up to 28 days of life or date of death from any cause, whichever came first.
  daily weight gain or loss of the participants in grams (g)
use of inotropes, plasma volume expanders and sodium bicarbonate therapy | Participants will be assessed for the use of inotropes, plasma volume expanders and sodium bicarbonate therapy from the date of randomization up to 28 days of life or date of death from any cause, whichever came first.
  total number of days participants required inotropic support
survival | up to 4 weeks
  participant survival or death

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No